CLINICAL TRIAL: NCT00415623
Title: A Double-Blind, Comparative Study Between Amlodipine 5mg And 10mg In Patients With Essential Hypertension For Whom Amlodipine 5mg Is Insufficiently Effective
Brief Title: A Comparative Study Between Amlodipine 10mg And 5mg With Hypertension For Whom 5mg Is Insufficient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0531085
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2008-12-09 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine 5mg (Active Comparator)
  Interventions: Drug: Amlodipine
- Amlodipine 10mg (Experimental)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 5mg/ day
  Arms: Amlodipine 5mg
Drug: Amlodipine — Amlodipine 10mg/ day
  Arms: Amlodipine 10mg

SUMMARY:
The changes in the trough systolic blood pressure from the baseline were assessed after 8 weeks of double-blind treatment with amlodipine 10 mg or amlodipine 5 mg

ELIGIBILITY:
Inclusion Criteria:

* Untreated Hypertensive Patients: An systolic blood pressure of >=160 mmHg or diastolic blood pressure >=100mmHg.
* Treated Hypertensive Patients: An systolic blood pressure of >=140 mmHg or diastolic blood pressure of >= 90 mmHg.
* Patients with insufficient response to 5 mg of amlodipine in the screening period:Two successive systolic blood pressure measurements at Visit 4 (Week -2) and Visit 5 (Week 0 = baseline) >=140 mmHg
* Patients with a screening treatment compliance rate >= 80%

Exclusion Criteria:

* Subjects with secondary hypertension (renal disease, pheochromocytoma, and Cushing's syndrome, etc.), severe hypertension (systolic blood pressure of 180 mmHg or higher, or diastolic blood pressure of 110 mmHg or higher), and malignant hypertension

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Japan (14):
  - Pfizer Investigational Site, Kasuya-gun, Fujuoka
  - Pfizer Investigational Site, Chikushino-shi, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Koga, Fukuoka
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Iruma, Saitama
  - Pfizer Investigational Site, Koshigaya, Saitama
  - Pfizer Investigational Site, Adachi-ku, Tokyo
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Meguro-ku, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Sumida City, Tokyo
  - Pfizer Investigational Site, Fukuoka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531085&StudyName=A%20Comparative%20Study%20Between%20Amlodipine%2010mg%20And%205mg%20With%20Hypertension%20For%20Whom%205mg%20Is%20Insufficient

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) centers in Japan
Pre-assignment Details: Consent was taken from 414 patients, 356 patients who met the screening criteria received amlodipine 5 mg. After the 8 weeks of screening treatment, patients who met the entry criteria for double-blind period were randomized to either the amlodipine 10 mg group or the amlodipine 5 mg group at a ratio of 1:1.
Groups:
- Amlodipine 5 mg: One amlodipine besilate 5 mg tablet and 1 amlodipine besilate 5 mg placebo tablet were administered once daily after breakfast for 8 weeks.
- Amlodipine 10 mg: Two amlodipine besilate 5 mg tablets were administered once daily after breakfast for 8 weeks.
Period: Overall Study
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Started | 154 | 151
Completed | 149 | 146
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 4
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg | Total
Number analyzed (Participants) | 154 | 151 | 305
Age, Customized [Number; unit: partcipants]
  < 20 years | 0 | 0 | 0
  20 to 44 years | 15 | 15 | 30
  45 to 64 years | 75 | 70 | 145
  >= 65 years | 64 | 66 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 59 | 129
  Male | 84 | 92 | 176
Region of Enrollment [Number; unit: participants]
  Japan | 154 | 151 | 305

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 8
Description: Mean change in the trough SBP
Time Frame: Baseline to Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
mmHg | -7.0 [-8.8 to -5.2] | -13.7 [-15.4 to -12.0]
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; The hypothesis of no group differences (null hypothesis) was tested against that of the amlodipine 10 mg arm being superior to the amlodipine 5 mg arm (alternative hypothesis). ANCOVA models with the trough SBP at baseline, body weight, and age as covariates, and the treatment group and study site as factors was used. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -6.7, 95% CI [-9.0 to -4.4]

2. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline to Week 8
Description: Mean change in the trough DBP
Time Frame: Baseline to Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
mmHg | -2.7 [-3.9 to -1.4] | -6.8 [-8.0 to -5.5]
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; The hypothesis of no group differences (null hypothesis) was tested against that of the amlodipine 10 mg arm being superior to the amlodipine 5 mg arm (alternative hypothesis). ANCOVA models with the trough DBP at baseline, body weight, and age as covariates, and the treatment group and study site as factors was used. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -4.1, 95% CI [-5.7 to -2.5]

3. Secondary Outcome: Combined Mean Change in SBP From Baseline to Week 6 and Week 8 (Mean by Patient)
Description: Arithmetic mean of Week 6 & Week 8 by patient for "Change from baseline in SBP at Week 6" and "Change from baseline in SBP at Week 8"
Time Frame: Baseline to Week 6 and Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
mmHg | -6.8 [-8.4 to -5.2] | -13.9 [-15.5 to -12.4]
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -7.1, 95% CI [-9.1 to -5.1]

4. Secondary Outcome: Combined Mean Change in DBP From Baseline to Week 6 and Week 8 (Mean by Patient)
Description: Arithmetic mean of Week 6 & Week 8 by patient for "Change from baseline in DBP at Week 6" and "Change from baseline in DBP at Week 8"
Time Frame: Baseline to Week 6 and Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
mmHg | -2.5 [-3.6 to -1.4] | -6.5 [-7.6 to -5.5]
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -4.0, 95% CI [-5.4 to -2.6]

5. Secondary Outcome: Number of Subjects Achieving the Target Blood Pressure Reduction Value at Week 8
Description: Target blood pressure reduction value based on Japan Society of Hypertension Guidelines for the Management of Hypertension 2004: SBP below 130 mmHg and DBP below 85 mmHg for <=64 years old; SBP below 140 mmHg and DBP below 90 mmHg for >=65 years old
Time Frame: Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
participants | 43 | 66
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; Proportions of participants (responder rates) were used for the statistical analyses. The hypothesis of no group differences (null hypothesis) was tested against that of the amlodipine 10 mg arm being superior to the amlodipine 5 mg arm (alternative hypothesis). The test was conducted based on a logistic regression model with baseline SBP value and body weight as covariates, and treatment group and age (<=64, >=65) as a factor. The significance level was 0.05 (two-sided); Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI [1.36 to 3.99]

6. Secondary Outcome: Combined Number of Subjects Achieving the Target Blood Pressure Reduction Value at Both Weeks 6 and 8
Description: as for outcome 5
Time Frame: Week 6 and Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
participants | 22 | 52
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.46, 95% CI [2.28 to 8.74]

7. Secondary Outcome: Number of Subjects Achieving the Target Blood Pressure Reduction Value and Whose SBP Decreased From Baseline by >= 10 mmHg at Week 8
Description: as for outcome 5
Time Frame: Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
participants | 35 | 61
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.55, 95% CI [1.50 to 4.36]

8. Secondary Outcome: Combined Number of Subjects Achieving the Target Blood Pressure Reduction Value and Whose SBP Decreased From Baseline by >= 10 mmHg at Both Weeks 6 and 8
Description: as for outcome 5
Time Frame: Week 6 and Week 8
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Amlodipine 5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 151 | 150
participants | 16 | 44
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Amlodipine 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.16, 95% CI [2.12 to 8.19]

9. Secondary Outcome: Trough Plasma Concentrations of Amlodipine -Amlodipine 5 mg
Time Frame: Baseline, Week 4 and Week 8
Population: Plasma concentration obtained after temporarily dosing discontinuation or not matched with the following conditions were excluded from the analysis; Steady-state condition: at least 80% drug compliance from the previous visit to the day of sampling; Trough condition: samples taken within ±10% of 24 hours from last dosing.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Baseline: After once daily administration of amlodipine 5 mg for 8 weeks in the screening period
Arm/Group | Baseline | Week 4 | Week 8
Number analyzed (Participants) | 147 | 146 | 145
ng/mL | 7.02 [6.5 to 7.5] | 6.83 [6.3 to 7.4] | 7.03 [6.6 to 7.5]

10. Secondary Outcome: Trough Plasma Concentrations of Amlodipine -Amlodipine 10 mg
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Baseline | Week 4 | Week 8
Number analyzed (Participants) | 145 | 144 | 143
ng/mL | 7.18 [6.7 to 7.7] | 16.9 [15.7 to 18.1] | 16.9 [15.7 to 18.2]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.